CLINICAL TRIAL: NCT06585618
Title: Multicenter Pediatric Deep Brain Stimulation Registry
Brief Title: A Multicenter Pediatric Deep Brain Stimulation Registry
Acronym: DBS-R
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Darius Ebrahimi-Fakhari, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00047069
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dystonia; Epilepsy in Children; Cerebral Palsy; Tourette Syndrome; Obsessive-Compulsive Disorder; Neurologic Disorder; Movement Disorders in Children; Movement Disorders; Deep Brain Stimulation
Keywords: Deep Brain Stimulation; DBS; movement disorder; movement disorders in children; dystonia; chorea; dyskinesia; epilepsy
MeSH Terms: conditions — Dystonia; Cerebral Palsy; Tourette Syndrome; Obsessive-Compulsive Disorder; Nervous System Diseases; Movement Disorders; Chorea; Dyskinesias; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is limited data on outcomes for children who have undergone deep brain stimulation (DBS) for movement disorders, and individual centers performing this surgery often lack sufficient cases to power research studies adequately. This study aims to develop a multicenter pediatric DBS registry that allows multiple sites to share clinical pediatric DBS data. The primary goals are to enable large-scale, well-powered analyses of the safety and efficacy of DBS in the pediatric population and to further explore and refine DBS as a therapeutic option for children with dystonia and other hyperkinetic movement disorders. Given the current scarcity of evidence available to clinicians, this centralized multicenter repository of clinical data is critical for addressing key research questions and improving clinical practice for pediatric DBS.

DETAILED DESCRIPTION:
The use of deep brain stimulation (DBS) has expanded to include multiple conditions in children including dystonia, epilepsy, Tourette syndrome and mood disorders. Despite its growing application, DBS remains a low-volume procedure in most pediatric centers, which limits opportunities for large-scale research studies. To overcome this challenge, an international data-sharing platform is essential for advancing knowledge about DBS in pediatric patients, particularly concerning surgical techniques and patient outcomes across various conditions.

This study aims to establish a multicenter pediatric DBS registry. With limited data on pediatric DBS outcomes and a small number of cases at individual centers, there is a need for a comprehensive registry to enable large-scale, well-powered analyses of DBS safety and effectiveness. The primary goals of this study are to:

* Establish and implement a multi-center pediatric DBS registry
* Facilitate large-scale analyses of DBS safety and effectiveness in children
* Refine DBS as a treatment option for dystonia and other hyperkinetic movement disorders in children.

Secondary objectives include:

* Identifying which patients benefit most from DBS
* Determining clinical variables that influence DBS responsiveness
* Identifying optimal implant sites for specific conditions
* Understanding the long-term effects of DBS in children
* Assessing the impact of DBS on the quality of life in pediatric patients

The study will involve both prospective and retrospective data collection from pediatric DBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients between ages of 0-18 years.
* Having received or scheduled to receive DBS for any neurological movement disorder.
* Parents or legal guardians are able to provide written consent for prospective enrollment.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of both female and male patients aged 0 to 18 years who have either received or are scheduled to receive deep brain stimulation (DBS) for any neurological disorder. Eligibility requires that parents or legal guardians are able to provide written consent for prospective enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Development of a Multi-Center Pediatric DBS Registry | 5 years
  This study will define DBS as a therapeutic option for children with dystonia, other hyperkinetic movement disorders, or epilepsy.

SECONDARY OUTCOMES:
Data Collection | 5 years
  Secondary objectives will focus on using the data collected to answer important research questions such as :
  1. Which patients benefit from DBS?
  2. Which clinical variables contribute to the responsiveness or nonresponsivness to DBS?
  3. Which implant sites are preferred?
  4. What are the long-term effects of DBS in the pediatric population?
  5. How does DBS affect quality of life in pediatric patients?

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Camfield P, Camfield C. Incidence, prevalence and aetiology of seizures and epilepsy in children. Epileptic Disord. 2015 Jun;17(2):117-23. doi: 10.1684/epd.2015.0736. PMID 25895502
- [Background] Zesiewicz TA, Sullivan KL, Hauser RA. Levodopa-induced dyskinesia in Parkinson's disease: epidemiology, etiology, and treatment. Curr Neurol Neurosci Rep. 2007 Jul;7(4):302-10. doi: 10.1007/s11910-007-0046-y. PMID 17618536
- [Background] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Background] Russ SA, Larson K, Halfon N. A national profile of childhood epilepsy and seizure disorder. Pediatrics. 2012 Feb;129(2):256-64. doi: 10.1542/peds.2010-1371. Epub 2012 Jan 23. PMID 22271699
- [Background] Sillanpaa M. Long-term outcome of epilepsy. Epileptic Disord. 2000 Jun;2(2):79-88. PMID 10954238
- [Background] Vasconcellos E, Wyllie E, Sullivan S, Stanford L, Bulacio J, Kotagal P, Bingaman W. Mental retardation in pediatric candidates for epilepsy surgery: the role of early seizure onset. Epilepsia. 2001 Feb;42(2):268-74. doi: 10.1046/j.1528-1157.2001.12200.x. PMID 11240601
- [Background] Wendorff J. [Epilepsy and mental retardation. The school's functioning in children with epilepsy]. Przegl Lek. 2010;67(11):1175-8. Polish. PMID 21442972
- [Background] Thompson R, Kerr M, Glynn M, Linehan C. Caring for a family member with intellectual disability and epilepsy: practical, social and emotional perspectives. Seizure. 2014 Nov;23(10):856-63. doi: 10.1016/j.seizure.2014.07.005. Epub 2014 Jul 19. PMID 25086700
- [Background] Sanger TD, Chen D, Fehlings DL, Hallett M, Lang AE, Mink JW, Singer HS, Alter K, Ben-Pazi H, Butler EE, Chen R, Collins A, Dayanidhi S, Forssberg H, Fowler E, Gilbert DL, Gorman SL, Gormley ME Jr, Jinnah HA, Kornblau B, Krosschell KJ, Lehman RK, MacKinnon C, Malanga CJ, Mesterman R, Michaels MB, Pearson TS, Rose J, Russman BS, Sternad D, Swoboda KJ, Valero-Cuevas F. Definition and classification of hyperkinetic movements in childhood. Mov Disord. 2010 Aug 15;25(11):1538-49. doi: 10.1002/mds.23088. PMID 20589866
- [Background] van Egmond ME, Kuiper A, Eggink H, Sinke RJ, Brouwer OF, Verschuuren-Bemelmans CC, Sival DA, Tijssen MA, de Koning TJ. Dystonia in children and adolescents: a systematic review and a new diagnostic algorithm. J Neurol Neurosurg Psychiatry. 2015 Jul;86(7):774-81. doi: 10.1136/jnnp-2014-309106. Epub 2014 Nov 13. PMID 25395479
- [Background] van Egmond ME, Lugtenberg CHA, Brouwer OF, Contarino MF, Fung VSC, Heiner-Fokkema MR, van Hilten JJ, van der Hout AH, Peall KJ, Sinke RJ, Roze E, Verschuuren-Bemelmans CC, Willemsen MA, Wolf NI, Tijssen MA, de Koning TJ. A post hoc study on gene panel analysis for the diagnosis of dystonia. Mov Disord. 2017 Apr;32(4):569-575. doi: 10.1002/mds.26937. Epub 2017 Feb 10. PMID 28186668
- [Background] Martin K, Jackson CF, Levy RG, Cooper PN. Ketogenic diet and other dietary treatments for epilepsy. Cochrane Database Syst Rev. 2016 Feb 9;2:CD001903. doi: 10.1002/14651858.CD001903.pub3. PMID 26859528
- [Background] Cunha JM, Carlini EA, Pereira AE, Ramos OL, Pimentel C, Gagliardi R, Sanvito WL, Lander N, Mechoulam R. Chronic administration of cannabidiol to healthy volunteers and epileptic patients. Pharmacology. 1980;21(3):175-85. doi: 10.1159/000137430. PMID 7413719
- [Background] Mechoulam R, Carlini EA. Toward drugs derived from cannabis. Naturwissenschaften. 1978 Apr;65(4):174-9. doi: 10.1007/BF00450585. PMID 351429
- [Background] Devinsky O, Marsh E, Friedman D, Thiele E, Laux L, Sullivan J, Miller I, Flamini R, Wilfong A, Filloux F, Wong M, Tilton N, Bruno P, Bluvstein J, Hedlund J, Kamens R, Maclean J, Nangia S, Singhal NS, Wilson CA, Patel A, Cilio MR. Cannabidiol in patients with treatment-resistant epilepsy: an open-label interventional trial. Lancet Neurol. 2016 Mar;15(3):270-8. doi: 10.1016/S1474-4422(15)00379-8. Epub 2015 Dec 24. PMID 26724101
- [Background] Fish DR, Smith SJ, Quesney LF, Andermann F, Rasmussen T. Surgical treatment of children with medically intractable frontal or temporal lobe epilepsy: results and highlights of 40 years' experience. Epilepsia. 1993 Mar-Apr;34(2):244-7. doi: 10.1111/j.1528-1157.1993.tb02405.x. PMID 8453932
- [Background] Paolicchi JM, Jayakar P, Dean P, Yaylali I, Morrison G, Prats A, Resnik T, Alvarez L, Duchowny M. Predictors of outcome in pediatric epilepsy surgery. Neurology. 2000 Feb 8;54(3):642-7. doi: 10.1212/wnl.54.3.642. PMID 10680797
- [Background] Wyllie E. Surgical treatment of epilepsy in pediatric patients. Can J Neurol Sci. 2000 May;27(2):106-10. PMID 10830341
- [Background] Harkness W. Temporal lobe resections. Childs Nerv Syst. 2006 Aug;22(8):936-44. doi: 10.1007/s00381-006-0140-5. Epub 2006 Jul 11. PMID 16832669
- [Background] Freitag H, Tuxhorn I. Cognitive function in preschool children after epilepsy surgery: rationale for early intervention. Epilepsia. 2005 Apr;46(4):561-7. doi: 10.1111/j.0013-9580.2005.03504.x. PMID 15816951
- [Background] Leiphart JW, Peacock WJ, Mathern GW. Lobar and multilobar resections for medically intractable pediatric epilepsy. Pediatr Neurosurg. 2001 Jun;34(6):311-8. doi: 10.1159/000056044. PMID 11455232
- [Background] Cossu M, Lo Russo G, Francione S, Mai R, Nobili L, Sartori I, Tassi L, Citterio A, Colombo N, Bramerio M, Galli C, Castana L, Cardinale F. Epilepsy surgery in children: results and predictors of outcome on seizures. Epilepsia. 2008 Jan;49(1):65-72. doi: 10.1111/j.1528-1167.2007.01207.x. Epub 2007 Jul 21. PMID 17645538
- [Background] Maehara T, Shimizu H, Kawai K, Shigetomo R, Tamagawa K, Yamada T, Inoue M. Postoperative development of children after hemispherotomy. Brain Dev. 2002 Apr;24(3):155-60. doi: 10.1016/s0387-7604(02)00010-4. PMID 11934511
- [Background] Shimizu H. Our experience with pediatric epilepsy surgery focusing on corpus callosotomy and hemispherotomy. Epilepsia. 2005;46 Suppl 1:30-1. doi: 10.1111/j.0013-9580.2005.461009.x. PMID 15816976
- [Background] Basheer SN, Connolly MB, Lautzenhiser A, Sherman EM, Hendson G, Steinbok P. Hemispheric surgery in children with refractory epilepsy: seizure outcome, complications, and adaptive function. Epilepsia. 2007 Jan;48(1):133-40. doi: 10.1111/j.1528-1167.2006.00909.x. PMID 17241220
- [Background] Gonzalez-Martinez JA, Gupta A, Kotagal P, Lachhwani D, Wyllie E, Luders HO, Bingaman WE. Hemispherectomy for catastrophic epilepsy in infants. Epilepsia. 2005 Sep;46(9):1518-25. doi: 10.1111/j.1528-1167.2005.53704.x. PMID 16146448
- [Background] Graham D, Tisdall MM, Gill D. Corpus callosotomy outcomes in pediatric patients: A systematic review. Epilepsia. 2016 Jul;57(7):1053-68. doi: 10.1111/epi.13408. Epub 2016 May 29. PMID 27237542
- [Background] Hallbook T, Lundgren J, Stjernqvist K, Blennow G, Stromblad LG, Rosen I. Vagus nerve stimulation in 15 children with therapy resistant epilepsy; its impact on cognition, quality of life, behaviour and mood. Seizure. 2005 Oct;14(7):504-13. doi: 10.1016/j.seizure.2005.08.007. Epub 2005 Sep 19. PMID 16176878
- [Background] Klinkenberg S, Majoie HJ, van der Heijden MM, Rijkers K, Leenen L, Aldenkamp AP. Vagus nerve stimulation has a positive effect on mood in patients with refractory epilepsy. Clin Neurol Neurosurg. 2012 May;114(4):336-40. doi: 10.1016/j.clineuro.2011.11.016. Epub 2011 Nov 30. PMID 22130047
- [Background] Klinkenberg S, van den Bosch CN, Majoie HJ, Aalbers MW, Leenen L, Hendriksen J, Cornips EM, Rijkers K, Vles JS, Aldenkamp AP. Behavioural and cognitive effects during vagus nerve stimulation in children with intractable epilepsy - a randomized controlled trial. Eur J Paediatr Neurol. 2013 Jan;17(1):82-90. doi: 10.1016/j.ejpn.2012.07.003. Epub 2012 Aug 9. PMID 22878130
- [Background] Terra VC, Furlanetti LL, Nunes AA, Thome U, Nisyiama MA, Sakamoto AC, Machado HR. Vagus nerve stimulation in pediatric patients: Is it really worthwhile? Epilepsy Behav. 2014 Feb;31:329-33. doi: 10.1016/j.yebeh.2013.10.011. Epub 2013 Nov 5. PMID 24210463
- [Background] Klinkenberg S, Aalbers MW, Vles JS, Cornips EM, Rijkers K, Leenen L, Kessels FG, Aldenkamp AP, Majoie M. Vagus nerve stimulation in children with intractable epilepsy: a randomized controlled trial. Dev Med Child Neurol. 2012 Sep;54(9):855-61. doi: 10.1111/j.1469-8749.2012.04305.x. Epub 2012 Apr 28. PMID 22540141
- [Background] Air EL, Ostrem JL, Sanger TD, Starr PA. Deep brain stimulation in children: experience and technical pearls. J Neurosurg Pediatr. 2011 Dec;8(6):566-74. doi: 10.3171/2011.8.PEDS11153. PMID 22132914
- [Background] Haridas A, Tagliati M, Osborn I, Isaias I, Gologorsky Y, Bressman SB, Weisz D, Alterman RL. Pallidal deep brain stimulation for primary dystonia in children. Neurosurgery. 2011 Mar;68(3):738-43; discussion 743. doi: 10.1227/NEU.0b013e3182077396. PMID 21164379
- [Background] Timmermann L, Pauls KA, Wieland K, Jech R, Kurlemann G, Sharma N, Gill SS, Haenggeli CA, Hayflick SJ, Hogarth P, Leenders KL, Limousin P, Malanga CJ, Moro E, Ostrem JL, Revilla FJ, Santens P, Schnitzler A, Tisch S, Valldeoriola F, Vesper J, Volkmann J, Woitalla D, Peker S. Dystonia in neurodegeneration with brain iron accumulation: outcome of bilateral pallidal stimulation. Brain. 2010 Mar;133(Pt 3):701-12. doi: 10.1093/brain/awq022. Epub 2010 Mar 5. PMID 20207700
- [Background] Borggraefe I, Mehrkens JH, Telegravciska M, Berweck S, Botzel K, Heinen F. Bilateral pallidal stimulation in children and adolescents with primary generalized dystonia--report of six patients and literature-based analysis of predictive outcomes variables. Brain Dev. 2010 Mar;32(3):223-8. doi: 10.1016/j.braindev.2009.03.010. Epub 2009 Apr 28. PMID 19403250
- [Background] Jinnah HA, Factor SA. Diagnosis and treatment of dystonia. Neurol Clin. 2015 Feb;33(1):77-100. doi: 10.1016/j.ncl.2014.09.002. PMID 25432724
- [Background] Anderson WS, Lenz FA. Surgery insight: Deep brain stimulation for movement disorders. Nat Clin Pract Neurol. 2006 Jun;2(6):310-20. doi: 10.1038/ncpneuro0193. PMID 16932575
- [Background] DeLong M, Wichmann T. Deep brain stimulation for movement and other neurologic disorders. Ann N Y Acad Sci. 2012 Aug;1265:1-8. doi: 10.1111/j.1749-6632.2012.06608.x. Epub 2012 Jul 23. PMID 22823512
- [Background] Yu H, Neimat JS. The treatment of movement disorders by deep brain stimulation. Neurotherapeutics. 2008 Jan;5(1):26-36. doi: 10.1016/j.nurt.2007.10.072. PMID 18164481
- [Background] Borggraefe I, Boetzel K, Boehmer J, Berweck S, Mueller-Felber W, Mueller K, Mehrkens JH, Heinen F. Return to participation - significant improvement after bilateral pallidal stimulation in rapidly progressive DYT-1 dystonia. Neuropediatrics. 2008 Aug;39(4):239-42. doi: 10.1055/s-0028-1112117. Epub 2009 Jan 22. PMID 19165713
- [Background] Fisher R, Salanova V, Witt T, Worth R, Henry T, Gross R, Oommen K, Osorio I, Nazzaro J, Labar D, Kaplitt M, Sperling M, Sandok E, Neal J, Handforth A, Stern J, DeSalles A, Chung S, Shetter A, Bergen D, Bakay R, Henderson J, French J, Baltuch G, Rosenfeld W, Youkilis A, Marks W, Garcia P, Barbaro N, Fountain N, Bazil C, Goodman R, McKhann G, Babu Krishnamurthy K, Papavassiliou S, Epstein C, Pollard J, Tonder L, Grebin J, Coffey R, Graves N; SANTE Study Group. Electrical stimulation of the anterior nucleus of thalamus for treatment of refractory epilepsy. Epilepsia. 2010 May;51(5):899-908. doi: 10.1111/j.1528-1167.2010.02536.x. Epub 2010 Mar 17. PMID 20331461
- [Background] Li MCH, Cook MJ. Deep brain stimulation for drug-resistant epilepsy. Epilepsia. 2018 Feb;59(2):273-290. doi: 10.1111/epi.13964. Epub 2017 Dec 7. PMID 29218702
- [Background] Coubes P, Echenne B, Roubertie A, Vayssiere N, Tuffery S, Humbertclaude V, Cambonie G, Claustres M, Frerebeau P. [Treatment of early-onset generalized dystonia by chronic bilateral stimulation of the internal globus pallidus. Apropos of a case]. Neurochirurgie. 1999 May;45(2):139-44. French. PMID 10448655
- [Background] Valentin A, Selway RP, Amarouche M, Mundil N, Ughratdar I, Ayoubian L, Martin-Lopez D, Kazi F, Dar T, Jimenez-Jimenez D, Hughes E, Alarcon G. Intracranial stimulation for children with epilepsy. Eur J Paediatr Neurol. 2017 Jan;21(1):223-231. doi: 10.1016/j.ejpn.2016.10.011. Epub 2016 Nov 1. PMID 27840024
- [Background] Marks WA, Honeycutt J, Acosta F, Reed M. Deep brain stimulation for pediatric movement disorders. Semin Pediatr Neurol. 2009 Jun;16(2):90-8. doi: 10.1016/j.spen.2009.04.001. PMID 19501337
- [Background] Lipsman N, Ellis M, Lozano AM. Current and future indications for deep brain stimulation in pediatric populations. Neurosurg Focus. 2010 Aug;29(2):E2. doi: 10.3171/2010.5.FOCUS1095. PMID 20672919
- [Background] Yan H, Toyota E, Anderson M, Abel TJ, Donner E, Kalia SK, Drake J, Rutka JT, Ibrahim GM. A systematic review of deep brain stimulation for the treatment of drug-resistant epilepsy in childhood. J Neurosurg Pediatr. 2019 Mar 1;23(3):274-284. doi: 10.3171/2018.9.PEDS18417. Epub 2018 Nov 30. PMID 30544364
- [Background] Fisher RS, Uematsu S, Krauss GL, Cysyk BJ, McPherson R, Lesser RP, Gordon B, Schwerdt P, Rise M. Placebo-controlled pilot study of centromedian thalamic stimulation in treatment of intractable seizures. Epilepsia. 1992 Sep-Oct;33(5):841-51. doi: 10.1111/j.1528-1157.1992.tb02192.x. PMID 1396427
- [Background] Kim SH, Lim SC, Yang DW, Cho JH, Son BC, Kim J, Hong SB, Shon YM. Thalamo-cortical network underlying deep brain stimulation of centromedian thalamic nuclei in intractable epilepsy: a multimodal imaging analysis. Neuropsychiatr Dis Treat. 2017 Oct 17;13:2607-2619. doi: 10.2147/NDT.S148617. eCollection 2017. PMID 29089767
- [Background] Valentin A, Garcia Navarrete E, Chelvarajah R, Torres C, Navas M, Vico L, Torres N, Pastor J, Selway R, Sola RG, Alarcon G. Deep brain stimulation of the centromedian thalamic nucleus for the treatment of generalized and frontal epilepsies. Epilepsia. 2013 Oct;54(10):1823-33. doi: 10.1111/epi.12352. Epub 2013 Sep 13. PMID 24032641
- [Background] Velasco AL, Velasco F, Jimenez F, Velasco M, Castro G, Carrillo-Ruiz JD, Fanghanel G, Boleaga B. Neuromodulation of the centromedian thalamic nuclei in the treatment of generalized seizures and the improvement of the quality of life in patients with Lennox-Gastaut syndrome. Epilepsia. 2006 Jul;47(7):1203-12. doi: 10.1111/j.1528-1167.2006.00593.x. PMID 16886984
- [Background] Velasco F, Velasco M, Jimenez F, Velasco AL, Brito F, Rise M, Carrillo-Ruiz JD. Predictors in the treatment of difficult-to-control seizures by electrical stimulation of the centromedian thalamic nucleus. Neurosurgery. 2000 Aug;47(2):295-304; discussion 304-5. doi: 10.1097/00006123-200008000-00007. PMID 10942002
- [Background] Velasco F, Velasco M, Ogarrio C, Fanghanel G. Electrical stimulation of the centromedian thalamic nucleus in the treatment of convulsive seizures: a preliminary report. Epilepsia. 1987 Jul-Aug;28(4):421-30. doi: 10.1111/j.1528-1157.1987.tb03668.x. PMID 3497802
- [Background] Lin JP, Lumsden DE, Gimeno H, Kaminska M. The impact and prognosis for dystonia in childhood including dystonic cerebral palsy: a clinical and demographic tertiary cohort study. J Neurol Neurosurg Psychiatry. 2014 Nov;85(11):1239-44. doi: 10.1136/jnnp-2013-307041. Epub 2014 Mar 3. PMID 24591458
- [Background] Keen JR, Przekop A, Olaya JE, Zouros A, Hsu FP. Deep brain stimulation for the treatment of childhood dystonic cerebral palsy. J Neurosurg Pediatr. 2014 Dec;14(6):585-93. doi: 10.3171/2014.8.PEDS141. Epub 2014 Oct 17. PMID 25325412
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] Lipsman N, Woodside DB, Giacobbe P, Hamani C, Carter JC, Norwood SJ, Sutandar K, Staab R, Elias G, Lyman CH, Smith GS, Lozano AM. Subcallosal cingulate deep brain stimulation for treatment-refractory anorexia nervosa: a phase 1 pilot trial. Lancet. 2013 Apr 20;381(9875):1361-1370. doi: 10.1016/S0140-6736(12)62188-6. Epub 2013 Mar 7. PMID 23473846
- [Background] Laxton AW, Tang-Wai DF, McAndrews MP, Zumsteg D, Wennberg R, Keren R, Wherrett J, Naglie G, Hamani C, Smith GS, Lozano AM. A phase I trial of deep brain stimulation of memory circuits in Alzheimer's disease. Ann Neurol. 2010 Oct;68(4):521-34. doi: 10.1002/ana.22089. PMID 20687206
- [Background] Andrade DM, Zumsteg D, Hamani C, Hodaie M, Sarkissian S, Lozano AM, Wennberg RA. Long-term follow-up of patients with thalamic deep brain stimulation for epilepsy. Neurology. 2006 May 23;66(10):1571-3. doi: 10.1212/01.wnl.0000206364.19772.39. Epub 2006 Mar 15. PMID 16540602
- [Background] Hung SW, Hamani C, Lozano AM, Poon YY, Piboolnurak P, Miyasaki JM, Lang AE, Dostrovsky JO, Hutchison WD, Moro E. Long-term outcome of bilateral pallidal deep brain stimulation for primary cervical dystonia. Neurology. 2007 Feb 6;68(6):457-9. doi: 10.1212/01.wnl.0000252932.71306.89. PMID 17283323
- [Background] Kumar R, Lozano AM, Montgomery E, Lang AE. Pallidotomy and deep brain stimulation of the pallidum and subthalamic nucleus in advanced Parkinson's disease. Mov Disord. 1998;13 Suppl 1:73-82. PMID 9613722
- [Background] Kumar R, Lozano AM, Sime E, Lang AE. Long-term follow-up of thalamic deep brain stimulation for essential and parkinsonian tremor. Neurology. 2003 Dec 9;61(11):1601-4. doi: 10.1212/01.wnl.0000096012.07360.1c. PMID 14663050
- [Background] Lozano AM, Mayberg HS, Giacobbe P, Hamani C, Craddock RC, Kennedy SH. Subcallosal cingulate gyrus deep brain stimulation for treatment-resistant depression. Biol Psychiatry. 2008 Sep 15;64(6):461-7. doi: 10.1016/j.biopsych.2008.05.034. Epub 2008 Jul 18. PMID 18639234
- [Background] Moro E, Lang AE, Strafella AP, Poon YY, Arango PM, Dagher A, Hutchison WD, Lozano AM. Bilateral globus pallidus stimulation for Huntington's disease. Ann Neurol. 2004 Aug;56(2):290-4. doi: 10.1002/ana.20183. PMID 15293283
- [Background] Moro E, Piboolnurak P, Arenovich T, Hung SW, Poon YY, Lozano AM. Pallidal stimulation in cervical dystonia: clinical implications of acute changes in stimulation parameters. Eur J Neurol. 2009 Apr;16(4):506-12. doi: 10.1111/j.1468-1331.2008.02520.x. PMID 19207733
- [Background] Moro E, Hamani C, Poon YY, Al-Khairallah T, Dostrovsky JO, Hutchison WD, Lozano AM. Unilateral pedunculopontine stimulation improves falls in Parkinson's disease. Brain. 2010 Jan;133(Pt 1):215-24. doi: 10.1093/brain/awp261. Epub 2009 Oct 21. PMID 19846583
- [Background] Rodriguez-Oroz MC, Obeso JA, Lang AE, Houeto JL, Pollak P, Rehncrona S, Kulisevsky J, Albanese A, Volkmann J, Hariz MI, Quinn NP, Speelman JD, Guridi J, Zamarbide I, Gironell A, Molet J, Pascual-Sedano B, Pidoux B, Bonnet AM, Agid Y, Xie J, Benabid AL, Lozano AM, Saint-Cyr J, Romito L, Contarino MF, Scerrati M, Fraix V, Van Blercom N. Bilateral deep brain stimulation in Parkinson's disease: a multicentre study with 4 years follow-up. Brain. 2005 Oct;128(Pt 10):2240-9. doi: 10.1093/brain/awh571. Epub 2005 Jun 23. PMID 15975946